CLINICAL TRIAL: NCT00647907
Title: An Open Label, Non-comparative, Multicenter Trial of the Efficacy, Safety and Toleration of Voriconazole in the Primary or Secondary Treatment of Invasive Fungal Infection
Brief Title: A Study of the Efficacy and Safety of Voriconazole for the Treatment of Fungal Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1501018
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Candidiasis; Cryptococcosis; Aspergillosis
MeSH Terms: conditions — Candidiasis; Cryptococcosis; Aspergillosis | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Oral or intravenous voriconazole. Oral tablets 400 mg twice daily loading dose on first day, followed by 200 mg twice daily taken at least 1 hour before or after a meal. Oral doses could be increased to a maximum of 300 mg twice daily if there was no clinical improvement after at least 3 days of treatment, no serious adverse events were reported, and clinical chemistry parameters were within the acceptable range for study entry. Intravenous treatment was initiated with a loading dose of 6 mg/kg twice daily for the first day followed by 4 mg/kg twice daily for at least 3 days (maximum infusion rate of 3 mg/kg/hr if administered by peripheral intravenous line). An intravenous loading dose was not required in patients who were restarted after oral treatment. Total duration of therapy (intravenous and oral) was 12 weeks.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Vfend for the treatment of fungal infections

ELIGIBILITY:
Inclusion Criteria:

* Systemic or invasive fungal infection
* Infection caused by organism for which there is no current treatment or infection with evidence of failure and/or intolerance to treatment with approved antifungal agents

Exclusion Criteria:

* Liver function test abnormalities
* Renal disease
* Fungal infections not considered to be invasive or systemic

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-04; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Serological response (evaluated by approved diagnostic serological tests [cryptococcosis, coccidiomycosis, and histoplasmosis]) at Weeks 2, 8, 12, and end of therapy. | Weeks 2, 8, 12, and end of therapy
Clinical response (evaluated based on change of attributable symptoms, signs, and/or bronchoscopic abnormalities present at baseline, judged by investigators, at Weeks 1, 2, 4, 8, 12, and end of therapy) at Weeks 1, 2, 4, 8, 12, and end of therapy. | Weeks 1, 2, 4, 8, 12 and end of therapy
Radiological response (evaluated based on all radiological abnormalities [X-ray, computed tomography scan] attributed to fungal infection compared to baseline) at Weeks 2, 8, 12, and end of therapy. | Weeks 2, 8, 12, and end of therapy
Mycological response (evaluated by the presences of fungal pathogen by relevant specimen [microscopy or histopathology]) at Weeks 2, 8, 12, and end of therapy. | Weeks 2, 8, 12, and end of therapy

SECONDARY OUTCOMES:
Global response to treatment (incorporating clinical, mycological, radiological, and serological responses as applicable) at end of therapy/Week 16. | End of therapy or Week 16
Change from baseline in laboratory parameters at Weeks 1, 2, 4, 8, 12, end of therapy, Week 16, and follow-up. | Weeks 1, 2, 4, 8, 12, end of therapy, Week 16, and follow-up
Change from baseline in electrocardiogram at Week 1 and end of therapy. | Week 1 and end of therapy
Incidence of adverse events at Weeks 1, 2, 4, 8, 12, end of therapy, Week 16, and follow-up. | Weeks 1, 2, 4, 8, 12, end of therapy, Week 16, and follow-up
Visual safety testing at Weeks 1, 8, 12, end of therapy, Week 16, and follow-up. | Weeks 1, 8, 12, end of therapy, Week 16, and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Taiwan (3):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501018&StudyName=A%20Study%20of%20the%20Efficacy%20and%20Safety%20of%20Voriconazole%20for%20the%20Treatment%20of%20Fungal%20Infections